CLINICAL TRIAL: NCT03849664
Title: A Multicentre Double-blind Placebo-controlled Randomized Study of Efficacy and Safety of Cytoflavin®, Intravenous Administration and Enteric-coated Tablets, Used in Elderly Patients for Prevention of Cognitive Decline After Major Surgery
Brief Title: Efficacy and Safety of Cytoflavin® Used in Elderly Patients for the Prevention of Cognitive Decline After Major Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CYT-COG-16
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Dysfunction
Keywords: postoperative cognitive decline
MeSH Terms: conditions — Cognitive Dysfunction; Postoperative Cognitive Complications | interventions — Inosine; Niacinamide; Riboflavin; Meglumine; Water; Povidone; stearic acid; Hypromellose Derivatives; Coloring Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cytoflavin® (Experimental): Patients of group I will receive the experimental drug Cytoflavin®, manufactured by POLYSAN (Russia), on the day before surgery, during the surgical intervention, and in the postoperative period. Cytoflavin® solution(Inosine + Nicotinamide + Riboflavin + Succinic Acid) will be administered IV for 7 days, and Cytoflavin® enteric-coated tablets (Inosine + Nicotinamide + Riboflavin + Succinic Acid) will be administered for 25 days (in total 32 days of treatment).
  Interventions: Drug: Cytoflavin® solution; Drug: Cytoflavin® enteric-coated tablet
- Placebo (Placebo Comparator): Patients of group II will receive placebo (manufactured by POLYSAN, Russia), on the day before surgery, during the surgical intervention, and in the postoperative period. Placebo solution will be administered IV for 7 days, and placebo enteric-coated tablets will be administered for 25 days (in total 32 days of treatment).
  Interventions: Drug: Placebo solution; Drug: Placebo enteric-coated tablet

INTERVENTIONS:
Drug: Cytoflavin® solution — Single drip infusion of 20 ml of Cytoflavin® solution in 200 ml of 0.9%NaCl intravenously once a day
  Other Names: Inosine + Nicotinamide + Riboflavin + Succinic Acid solution
  Arms: Cytoflavin®
Drug: Cytoflavin® enteric-coated tablet — 2 tablets, orally, with 100 ml of drinking water, 30 minutes before meals, 2 times a day, with an interval of 8-10 hours (but no later than 18:00).
  Other Names: Inosine+Nicotinamide+Riboflavin+Succinic Acid tablet
  Arms: Cytoflavin®
Drug: Placebo solution — Single drip infusion of 20 ml of placebo solution in 200 ml of 0.9%NaCl intravenously once a day
  Other Names: riboflavin; meglumine, soduim hydroxide, water
  Arms: Placebo
Drug: Placebo enteric-coated tablet — 2 tablets, orally, with 100 ml of drinking water, 30 minutes before meals, 2 times a day, with an interval of 8-10 hours (but no later than 18:00).
  Other Names: povidone, calcium stearate, hypromellose, polysorban, dyes
  Arms: Placebo

SUMMARY:
Postoperative cognitive impairment develops in the early and continues in the late postoperative period; it is manifested by impaired memory, attention, concentration and other higher cortical functions (thinking, speech). Early studies demonstrated the positive impact of perioperative administration of Cytoflavin (Inosine + Nicotinamide + Riboflavin + Succinic Acid), which prevented impairments of intelligence, speech, and attention after cardiac surgery, both in conditions of cardiopulmonary bypass and on a working heart. The aim of the present study is to evaluate the safety and efficacy of Cytoflavin for the prevention of cognitive disorders after major surgeries performed in elderly patients.

DETAILED DESCRIPTION:
Cytoflavin® (Inosine + Nicotinamide + Riboflavin + Succinic Acid) is a combination drug, which improves coronary and cerebral blood flow, activates metabolic processes in the central nervous system, restores impaired consciousness, promotes regression of neurological symptoms and improvement of cognitive functions of the brain. It has a quick awakening effect in post-anesthetic depression of consciousness. The positive effect of Cytoflavin® on cognitive function has been previously shown in patients with dyscirculatory encephalopathy and acute stroke, as well as in a population of patients during cardiac surgery in cardiopulmonary bypass and working heart. The present study aims to evaluate the opportunity of prevention of postoperative cognitive decline by administration of Cytoflavin® at a sequential regimen, starting from intravenous infusions and followed by oral intake during 1 month.

Study objectives:

1. To study the efficacy of Cytoflavin® administered in elderly patients age for the prevention of cognitive decline after major surgery.
2. To study the safety and tolerability of Cytoflavin® in elderly patients for after major surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Men and women aged 60-80 years, inclusive.
3. Planned cardiac surgery, which does not assume the use of a cardiopulmonary bypass.
4. Planned or delayed orthopedic surgery (hip joint endoprosthetics, osteosynthesis for fractures of the proximal third of the hip, etc.), under general or combined anesthesia.
5. Legal capacity of the patient
6. Absence of dementia (MoCA≥17, MMSE≥19)
7. Lack of reproductive potential or
8. Consent to use adequate methods of contraception

Exclusion Criteria:

1. Hypersensitivity to any component of the study drug
2. Emergency surgery
3. Repeated surgery or reoperation
4. Anesthesia risk ASA≥5
5. Severe visual or hearing impairment which impedes the performance of neuropsychological tests
6. Operation under general anesthesia in the previous 3 months
7. Severe renal failure requiring replacement of renal function (dialysis)
8. Severe hepatic failure (class C and above in Child-Pugh)
9. Chronic obstructive pulmonary disease
10. Terminal stage of other chronic incurable diseases
11. Decompensated diabetes
12. A history of oncological diseases, mental illness, HIV infection, syphilis, tuberculosis, alcohol or drug addiction
13. The use of 5 or more units of alcohol per week in the previous 3 months
14. Diagnosis of mental or neurodegenerative disease (e.g. schizophrenia, Parkinson's disease, clinically manifest depression)
15. Permanent intake of psychotropic drugs (neuroleptics, tranquilizers, antidepressants)
16. Course intake of nootropic drugs in the previous 3 months
17. Communicative, sensory, motor, or any other deficiency that does not allow the patient to adequately assess their behavior and correctly fulfill the conditions of the study protocol.
18. The presence in the history of any significant, according to the physician-researcher, condition that prevents the inclusion of the patient in the study.
19. Participation in any clinical study in the previous 3 months
20. Employees of the study centres and their family members.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) scale score | 32 days
  The MoCA test is a one-page 30-point test, ranging between 0 and 30, where 0 is the worst and 30 is the best result; a score of 26-30 or over is considered to be normal. Outcome measure is the change in the MoCA scale score by the end of the treatment course compared with the preoperative score.

SECONDARY OUTCOMES:
The Mini-Mental State Examination (MMSE) scale | 32 days
  MMSE test is a 30-point questionnaire; any score greater than or equal to 24 points (out of 30) indicates a normal cognition; below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. Outcome measure will be the change of MMSE scale score by the end of the treatment course compared to the preoperative score
The Mini-Mental State Examination (MMSE) follow-up score | 90 days
  MMSE test is a 30-point questionnaire; any score greater than or equal to 24 points (out of 30) indicates a normal cognition; below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. Outcome measure will be the change of MMSE scale score by the end of the follow-up period
Montreal Cognitive Assessment (MoCA) follow-up | 90 days
  The MoCA test is a one-page 30-point test, ranging between 0 and 30, where 0 is the worst and 30 is the best result; a score of 26-30 or over is considered to be normal. Outcome measure is the change of the MoCA scale score by the end of the follow-up period
Median group Mini-Mental State Examination (MMSE) score | day 7, 32, 90
  MMSE test is a 30-point questionnaire; any score greater than or equal to 24 points (out of 30) indicates a normal cognition; below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. Outcome measure will be the difference between median group total scores on the MMSE scale.
Median Montreal Cognitive Assessment (MoCA) scale score | day 7, 32, 90
  The MoCA test is a one-page 30-point test, ranging between 0 and 30, where 0 is the worst and 30 is the best result; a score of 26-30 or over is considered to be normal. Outcome measure is the difference in median group values of the MOCA scale
Proportion of postoperative delirium | day 3-6
  The proportion of patients who developed postoperative delirium in the first 96 hours after surgery according to the results of CAM-ICU
Length of stay in the ICU | day 32
  Length of stay in the ICU
Mortality | day 32
  Mortality in the postoperative period in the experimental and control groups
Postoperative cognitive decline | day 32, day 90
  The proportion of patients with a decrease in the results of two or more neuropsychological tests by more than 20% by the end of the treatment course and by the end of the follow-up period compared the baseline values
Quality of life score | day 90
  Change in the overall score for the EQ-5D questionnaire for assessing the quality of life
Independence and activity | day 32
  The proportion of patients dependent in at least two daily functions according to the results of the Katz Daily Activity Index at the end of the treatment course
Anxiety/depression | day 32, day 90
  The group average score by Hospital Anxiety and Depression Scale (HADS) at the end of the treatment course and at the end of the follow-up period. The HADS is a fourteen item scale, a person can score between 0 and 21 for either anxiety or depression, where scores on each scale can be interpreted in ranges: normal (0-7), mild (8-10), moderate (11-14) and severe (15-21).

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana V Kharitonova, MD, PhD, Study Director — St. Petersburg Research Institute of Emergency Medicine n.a. I.I. Dzhanelidze
Locations (13):
- Russia (13):
  - Regional Clinical Hospital № 3, Chelyabinsk
  - Central Clinical Hospital with a polyclinic of the Office of the President of the Russian Federation, Moscow
  - Alexandrovskaya City Hospital, Saint Petersburg
  - City Hospital №15, Saint Petersburg
  - City Hospital №38 named after N.A. Semashko, Saint Petersburg
  - City Hospital №40 of the Kurortny District, Saint Petersburg
  - Hospital for War Veterans, Saint Petersburg
  - I. P. Pavlov 1st St. Petersburg State Medical University, Saint Petersburg
  - Military Medical Academy named after S.M. Kirov, Saint Petersburg
  - Pokrovskaya City Hospital, Saint Petersburg
  - GBUZ YAO "Regional Clinical Hospital", Yaroslavl
  - Research center of specialized types of medical care "Ural Institute of Cardiology", Yekaterinburg
  - Ural State Medical University, Yekaterinburg

REFERENCES:
- [Background] Kovalenko A.L., Nagibovich O.A., Vishnevsky A.Yu., Belekhov G.A., Gubaidullin R.R., Popov D.V., Agafiina A.S. Use of a Neurometabolism-Targeting Drug in Prevention of Postoperative Cognitive Dysfunction. General Reanimatology. 2022;18(2):12-21. https://doi.org/10.15360/1813-9779-2022-2-12-21
- See also: Related Info — https://doi.org/10.15360/1813-9779-2022-2-12-21